CLINICAL TRIAL: NCT02116556
Title: Effects of Rifaximin Treatment in Patients With Acute Alcoholic Hepatitis: A Comparative Pilot Study
Brief Title: Effects of Rifaximin in Patients With Acute Alcoholic Hepatitis
Acronym: RIFA-AAH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Germans Trias i Pujol Hospital (Other); Hospital del Mar (Other); Hospital de Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIFA-AAH.
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Alcoholic Hepatitis
Keywords: Alcoholic Hepatitis; Bacterial Infections; Acute-on-Chronic Liver Failure
MeSH Terms: conditions — Hepatitis, Alcoholic; Bacterial Infections; Acute-On-Chronic Liver Failure | interventions — Prednisone; Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisone (Active Comparator): Prednisone PO 40mg/day for 30 days plus standard supportive care measurements
  Interventions: Drug: Prednisone
- Prednisone plus Rifaximin (Experimental): Prednisone PO 40mg/day for 30 days plus Rifaximin PO 1200 mg/day for 90 days plus standard supportive care measurements
  Interventions: Drug: Prednisone; Drug: Rifaximin

INTERVENTIONS:
Drug: Prednisone — Prednisone PO 40mg/day or IV equivalent dosage for 30 days. Patients not responding at 7 days (e.g. Lille Model ≥ 0.45) treatment with Prednisone will be suspended.
Drug: Rifaximin — Rifaximin PO 1200 mg/day for 90 days
  Arms: Prednisone plus Rifaximin

SUMMARY:
Acute alcoholic hepatitis (AAH) is a serious condition and one of the most frequent causes of Acute-on-Chronic Liver Failure. The current standard therapy (corticosteroids) is theme of debate and unsatisfactory in many patients (year mortality: 30%). One of the main causes of death is bacterial infections, which affect 40-50% of patients at 90 days. Intestinal decontamination with rifaximin (a nonabsorbable antibiotic) reduces endotoxemia, improves liver function and reduces the complications of decompensated alcoholic cirrhosis.

The Hypothesis/Objective: To assess whether oral decontamination with rifaximin prevents the development of infections associated with AAH and analyze its consequences.

DETAILED DESCRIPTION:
Design: Open multicenter comparative study. A cohort (n = 66) will receive rifaximin (1200 mg / d) for 90 days. Results will be compared with those of a cohort of AAH prospectively included in an observational study. Both groups with a uniform treatment protocol (which includes the administration of corticosteroids and standardized treatment for complications of liver failure). Patients will be monitorized until hospital discharge and a follow-up visit at 7, 30, 45, 60 and 90 days will be performed.

Endpoints:

1. Primary endpoint: Bacterial infections after 90 days.
2. Secondary endpoints: :

2.1. Liver function tests 2.2. Levels of endotoxemia 2.3. Complications of liver cirrhosis. 2.4. Survival

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 and <70 years of age.
* Active alcohol abuse and excessive alcohol consumption prior to admission defined as > 50 g per day for men and> 40 g per day for women.
* Jaundice (Bilirubin >2 mg/dl) for no more than 3 months.
* Clinical suspicion of Alcoholic Hepatitis with a modified Maddrey's Discriminant Function > 32 points.

Exclusion Criteria:

* Hypersensitivity to Rifaximin
* Advanced Chronic or Terminal illness. Advanced Chronic illness will be defined as: all conditions evolved into a clinical stage to limit the patient's functional status (eg, heart failure NYHA> II, COPD PCO2> 50 mmHg or PO2 <60 mmHg, stroke or other disabling neurological disease, disabling or uncontrolled oncological conditions, etc ...).

Terminal illness will be defined as any clinical conditions with a survival expectancy less than 3 months

* Hepatocellular carcinoma (previously diagnosed) beyond Milan's criteria.
* Complete portal vein thrombosis (previously diagnosed).
* Autoimmune liver disease.
* Hepatitis B and C and HIV infection (anti-HCV, surface HBV antigen and anti-HIV positive).
* Pregnancy or nursing.
* Use of Rifaximin during the previous 2 months.
* Treatment with Pentoxifylline.
* Lack of informed consent.

Removal criteria:

* Lack of histological confirmation of Alcoholic Hepatitis during the first 7 days after inclusion.

Because there are no non-diagnostic tools to diagnose alcoholic hepatitis, histological confirmation is required in all patients (preferably through a transjugular biopsy): alcoholic hepatitis will be diagnosed on the presence of the following histologic features:

Hepatocellular damage (eg, hepatocyte ballooning and presence of Mallory-Denk bodies).

Inflammatory infiltrate (predominantly polymorphonuclear cells). Pericellular or sinusoidal fibrosis.

* Hepatocellular carcinoma beyond Milan's criteria diagnosed during the first 7 days after inclusion.
* Complete portal vein thrombosis diagnosed during the first 7 days after inclusion.
* Protocol violation.
* Severe adverse event directly related with Rifaximin.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Rate of bacterial infections | 90 days
  Development of any bacterial infection.

SECONDARY OUTCOMES:
Rate of Decompensations of Liver Cirrhosis | 90 days
  Development of any liver cirrhosis decompensations
  1. Hepatic Encephalopathy
  2. Acute Kidney Injury (including Hepatorenal Syndrome)
  3. Acute variceal bleeding
  4. Ascites
  5. Death

OTHER OUTCOMES:
Endotoxemia serum levels | 90 days
  Measurement of serum changes in endotoxemia levels during the rifaximin treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Vargas, MD, Principal Investigator — Internal Medicine Service. Vall d'Hebron Hospital
Locations (4):
- Spain (4):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Vall d'Hebron Hospital, Barcelona